CLINICAL TRIAL: NCT04995874
Title: Supplementation Trial of KOKO Plus Among HIV Exposed Children in Accra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noguchi Memorial Institute for Medical Research (Other)
Collaborators: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021X018.NMI
Record Dates: First submitted 2021-08-06; First posted 2021-08-09 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-08

CONDITIONS: HIV Infections; Nutrition Poor; Child Development
Keywords: HIV-Exposed; Nutrient Status; KOKOPlus
MeSH Terms: conditions — HIV Infections; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): KOKOPlus protein and micronutrient powder , a complementary food supplement containing soya powder, sugar and oil along with the essential amino acid lysine and a micronutrient mix was formulated. Two weeks' supply of KOKOPlus sachets will be given to intervention arm participants every fortnight for 6 months to be mixed into any cereal, soup, stew, or other food given to the children.
  Interventions: Dietary Supplement: KOKOPlus protein and micronutrient powder
- Control (No Intervention): This arm will receive no supplement and no placebo for the duration of the study.,

INTERVENTIONS:
Dietary Supplement: KOKOPlus protein and micronutrient powder — KokoPlus, a complementary food supplement was formulated by using linear programming methodology to improve the protein quality as well as the micronutrient and macronutrient content of commonly consumed traditional complementary (baby) foods in Ghana . It contains soya powder, sugar and oil along with the essential amino acid lysine and a micronutrient mix. It complies with WHO's complementary feeding guidelines, FAO/WHO recommended micronutrient intake (RNI) and the WHO's guidelines for protein and essential amino acid intake for children in the age group of 6 to 24 months. A daily supply of KokoPlus achieves 30% of the total recommended energy, 60% of total protein and 40% of total fat requirements from complementary foods. It also meets 35-55% of minimum intake of essential amino acids and 50-150% RNI based on the total daily requirements.
  Arms: Intervention

SUMMARY:
The overall aim of the research is to conduct a randomised controlled trial of KOKOPlus in young HIV exposed children attending HIV clinics in Accra, Ghana to test the effectiveness of KOKOPlus over a period of 6 months to improve nutritional status and child development in HIV exposed children 6-18 months of age in Accra

DETAILED DESCRIPTION:
The specific objectives are to accomplish the following

1. To test the effectiveness of KOKOPlus to improve the nutritional status of HIV exposed infants aged 6-18 months.
2. To measure and compare nutritional status in intervention and control arms by monitoring growth in terms of height and weight over the period of 6 months
3. To measure and compare micronutrient status of intervention and control arms by comparing baseline midline and endline measurements of hemoglobin levels.
4. To measure and compare morbidity rates of intervention and control arms.
5. To measure and compare rates of achievement of child development goals between intervention and control arms using a standardized tool, the Caregiver Reported Early Development Instrument (CREDI).
6. To understand and record experiences relating to the use of KOKOPlus of mothers/caregivers in the intervention arm through focus group discussion

ELIGIBILITY:
Inclusion Criteria:

* Mother-infant dyads; HIV positive mothers and children between 6 and 12 months of age attending antiretroviral (ART) Clinics and child HIV Clinics.

Exclusion Criteria:

* Mothers who decline to participate in the study

Children with severe acute malnutrition (mid-upper arm circumference <115 mm or a weight-for-height/length <-3 Z-scores of the WHO growth standards).

Children on hospital admission

Children with diagnosed or apparent congenital conditions such as encephalitis, cleft palate, hole in heart, which negatively affect the child's ability to eat and/or growth.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 649 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-06-25 (Estimated)

PRIMARY OUTCOMES:
Anthropometry | 6 months
  Length-for-age Z score, Weight-for-age Z score. Weight for length Z score
Haemoglobin | 6 months
  (g/dl), anaemia
Child developmental Milestones achieved | 6 months

SECONDARY OUTCOMES:
Morbidity | 6 months
  Incidence of fever, malaise, loss of appetite

CONTACTS AND LOCATIONS:
Overall Officials: Gloria K Folson, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (6):
- Ghana (6):
  - 37 Military Hospital, Accra, Greater Accra Region
  - Greater Accra Regional Hospital, Accra, Greater Accra Region
  - Korle-bu Teaching Hospital, Accra, Greater Accra Region
  - Princess Marie Louise Children's Hospital, Accra, Greater Accra Region
  - Ashaiman Polyclinic, Ashaiman, Greater Accra Region
  - Tema General Hospital, Tema, Greater Accra Region

IPD SHARING:
Plan to Share IPD: No